CLINICAL TRIAL: NCT01938690
Title: Effect of Transcranial Magnetic Stimulation on Motor Recovery of Upper Limb Among Stroke Survivors: Pilot Study
Brief Title: Effect of Transcranial Magnetic Stimulation on Recovery of Upper Limb Among Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, A. M. Barrett, MD, Director Stroke Lab, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-758-12
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Stroke
Keywords: stroke, transcranial magnetic stimulation, rehabilitation
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham stimulation (Sham Comparator): Sham stimulation on the scalp of unaffected brain
  Interventions: Device: Transcranial magnetic stimulation (TMS)
- transcranial magnetic stimulation (Experimental): transcranial magnetic stimulation on unaffected brain
  Interventions: Device: Transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Device: Transcranial magnetic stimulation (TMS) — 8 sessions of TMS followed by task specific training

SUMMARY:
Approximately two thirds of stroke survivors have profoundly impaired function of the upper limb. Currently the main stay of the treatment for upper limb motor function is rehabilitation therapy focusing on repetitive and skillful task practice (task-oriented therapy) which has been shown to induce substantial functional reorganization in the undamaged motor cortex and functional recovery. In spite of rehabilitation therapy, functional recovery of arm and hand function is limited to one third of stroke survivors and there is a great need for adjunct treatment to current practice. Repetitive Transcranial Magnetic Stimulation (rTMS) is a noninvasive means of stimulating nerve cells in superficial areas of the brain and emerging as a novel method of modulating cortical excitability and promoting functional recovery after stroke. There have been studies using rTMS to improve motor function after stroke. However, whether 1Hz rTMS can enhance the effect of the task-oriented therapy on upper limb function after stroke has not been investigated. In this pilot proposal, we intend to investigate the feasibility of 1Hz rTMS on unaffected hemisphere as an adjunct to task-oriented therapy to improve upper limb motor function among stroke patients. The information obtained from this pilot study will provide a platform for the future randomized control trials combining the rTMS and task-oriented therapy to enhance motor recovery among stroke survivors.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

--≥18 years of age

* Ability to give informed consent
* An unilateral ischemic stroke of onset 6-36 months prior to the study
* No other known brain abnormalities by medical history or by MRI
* Affected upper limb function of score 2-6 in Chedoke Arm and Hand Inventory
* Enrolled or planned to be enrolled in occupational therapy at Kessler Institute for Rehabilitation as an outpatient

Exclusion Criteria:

* More than one stroke (Transient Ischemic Attack not a reason for exclusion) Neurological conditions other than stroke (brain tumor, Parkinson's disease, etc)
* History of epilepsy or unprovoked seizures
* Family history of epilepsy (father, mother, children, siblings with diagnosis of epilepsy)
* Implanted medical devices (pacemakers, defibrillators, medical pump, implanted brain stimulator, aneurysm clip, carotid or cerebral stents, central venous catheter, cochlear implant, internal hearing aids)
* Damaged skin or skull of head
* Excessive spasticity of upper limb as indicated by Modified Ashworth Spasticity Scale >2/4
* Recent injection of antispastic medications (Botulinum toxin, phenol) of the last 3 months or scheduled such injection during the study period
* Severe sensory deficits as measured by a score of 2 on item 8 of the National Institute of Health (NIH) stroke scale
* Severe aphasia as measured by a score of ≥2 on item 9 of NIH stroke scale
* Being determined to be medically unstable by a physician
* Being pregnant or trying to become pregnant
* Past or current alcohol abuse, illicit drug use, or significant mental illness (schizophrenia, major depression, manic disorders)
* Working with metal currently or in the past
* Tattoo with metal based ink on the head or neck
* Unable to answer the questionnaires in the consent form correctly

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Upper limb function (Fugl Meyer score) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: A.M. Barrett, MD, Study Director — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States